CLINICAL TRIAL: NCT06230341
Title: Patient Safety Incidents in Coordinated Primary Care Teams: a Multi-method Study
Acronym: EVIDENS-Prim
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Université de Nantes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC23_0402; RSP22N005 (Other Grant/Funding Number: French Ministry of Health: Direction générale offre de soins)
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Adverse Event
Keywords: Healthcare; Adverse event; Safety culture; Patient safety; Learning
MeSH Terms: interventions — Health Services Research

STUDY DESIGN:
Intervention Model Description: Descriptive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Learning system benefits MSPs (Experimental): MSPs benefit from a learning system (described in the intervention section). MSPs are encouraged to report PSIs through the web platform provided after the initial training in each MSP and during the period of methodological support.
  Interventions: Other: Health Services Research

INTERVENTIONS:
Other: Health Services Research — MSPs benefit from a learning system. The learning system combines an individualised support programme provided by a regional support structure for quality and safety in health care (QualiREL Santé) and the provision of a web platform. Based on the 4 dimensions of the Shortell model, the support programme includes initial training (6 months) and personalised methodological support (18 months) for each MSP. A web platform is provided to MSPs to enable them to implement the full approach of the Risk Management Support Programme. It provides support for reporting, analysis and management of PSIs.

SUMMARY:
In France, improving the practice of health professionals working in coordinated primary care teams (health centres called Maisons de Santé Pluriprofessionnelles - MSPs) could be facilitated by a learning system consisting of (i) a risk management support programme and (ii) the provision of a comprehensive online system combining training, reporting and support for the analysis and management of patient safety incidents (PSIs).

EVIDENS-Prim is a multi-method, multi-centre, prospective study. It aims to describe the PSIs that occur in MSPs, using an international classification system, and to describe the ways in which professionals have adopted a global approach to PSIs management, from PSI reporting to feedback.

DETAILED DESCRIPTION:
This method combines:

- (i) A sequential study of PSIs analysis. The sequential study will take place in three stages (coder training, collection of PSIs data via the web platform, PSIs coding).

Each PSIs reported by professionals during the implementation of the risk management support programme will be coded using the PISA multi-axial classification system (based on the WHO's International Classification for Patient Safety in Primary Care). These codes will be used to describe PSIs in coordinated practice.

- (ii) An implementation study of the learning system. The learning system is described in the intervention section. During the implementation study, two types of data collection (quantitative and qualitative) will be mobilised at the end of the support to the QualiREL Santé Regional Support Structure.

The main objective of the study is:

- To Describe PSIs occurring in MSPs as part of the coordinated exercise and over an 18-month period, according to the 4 coding frameworks of the PISA classification: (i) types of events (main and contributing), (ii) contributing factors, (iii) outcomes of PSIs, (iv) severity of harm.

The secondary objectives, linked to the evaluation of the implementation of the learning system, are

* To examine the acceptance of the learning system by the teams,
* To describe the effective use of the web platform by professionals,
* To describe the MSP's ownership of the risk management support programme.

ELIGIBILITY:
Inclusion Criteria:

* Characteristics of the MSPs included in the study:
* Located in the Pays de la Loire region;
* Having a contract with a health insurance (specifications and financing defined nationally) for at least 1 year;
* Agreeing to take part in the project;
* Having a quality representative or committing to appoint one when they join the project.

Characteristics of professionals working in MSPs included:

* All independent health professionals involved in the MSP: general practitioners and, depending on the MSP, nurses, pharmacists, podiatrists, physiotherapists, midwives, speech therapists, dentists, occupational therapists, psychomotor therapists, etc,)
* All professionals involved in MSP outside the health sector: (coordinators, medical assistants, independent psychologists, etc.),
* agree to take part in the project.

Exclusion Criteria:

Other group exercise modalities or other forms of coordinated exercise (other than MSP) do not have a quality representative on their team and will not be considered for inclusion.

Characteristics of MSPs not included in the research:

- Where the members of the research team work.

Characteristics of professionals working in MSPs included:

- Not included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of PSIs occurring in MSPs according to the 4 coding frameworks of the PISA classification: 1-by type | PSIs reported by MSP professionals in the 18 months following the initial training provided
  Repartition, according to the PISA classification, of PSIs reported by MSP professionals in the 18 months following the initial training provided, by type: the number of PSIs for each type out of the total number of PSIs reported.
Distribution of PSIs occurring in MSPs according to the 4 coding frameworks of the PISA classification: 2- by contributing factors | 18 months
  Repartition, according to the PISA classification, of PSIs reported by MSP professionals in the 18 months following the initial training provided, by contributing factors : number of PSIs for each contributing factor (e.g. factors related to the patient, staff, equipment, organisation, etc.) out of the total number of PSIs reported.
Distribution of PSIs occurring in MSPs according to the 4 coding frameworks of the PISA classification: 3-by results | 18 months
  Repartition, according to the PISA classification, of PSIs reported by MSP professionals in the 18 months following the initial training provided, by results: number of PSIs for each result (no harm, clinical harm, team harm) out of the total number of PSIs reported.
Distribution of PSIs occurring in MSPs according to the 4 coding frameworks of the PISA classification: 4-by severity | 18 months
  Repartition, according to the PISA classification, of PSIs reported by MSP professionals in the 18 months following the initial training provided, by severity: number of PSIs of each severity (e.g. no harm, mild, moderate or severe harm, death) out of the total number of PSIs reported.

SECONDARY OUTCOMES:
Description of MSP professionals' acceptance of learning system | 3 months
  Analysis of the main themes and sub-themes of the acceptability of the learning system from the semi-directed interviews and focus groups conducted with MSP professionals.
Description of the behaviour of users of the online system in the 18 months following the provision of initial training | 18 months
  Export from the web platform of
  * the number of professionals who have validated the opening of their account on the web platform,
  * the number of professionals who have declared at least one PSI,
  * the number of modifications made to the PSIs declaration,
  * the number of declarations in anonymous mode,
  * the number of updates of action sheets corresponding to improvement actions.
Description of the MSP's behaviour in implementing the risk management support programme during the 18 months following the provision of the initial training. | 18 months
  Description: Export from the web platform of
  * the number of PSI declarations
  * the number of systemic analyses of PSIs carried out,
  * the number of types of contributing factors identified by the analysis (variable categories defined according to the analysis methods),
  * the number of analyses identifying security barriers (by type: present and effective / present and ineffective / absent),
  * the number of improvement actions planned / completed / abandoned.

IPD SHARING:
Plan to Share IPD: No